CLINICAL TRIAL: NCT02129101
Title: Phase I/Ib Study of Azacitidine or Decitabine With Hedgehog Pathway Inhibition in Myeloid Malignancies
Brief Title: Azacitidine and Sonidegib or Decitabine in Treating Patients With Myeloid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1389; NCI-2014-00866 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Mod13-009003-08; MC1389 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-08

CONDITIONS: Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndrome; Essential Thrombocythemia; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm; Polycythemia Vera; Previously Treated Myelodysplastic Syndrome; Primary Myelofibrosis; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Polycythemia Vera; Primary Myelofibrosis; Leukemia, Myeloid, Acute | interventions — Azacitidine; Decitabine; Injections; sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (azacitidine, sonidegib, decitabine) (Experimental): Patients receive azacitidine SC or IV on days 1-7, sonidegib PO QD on days 1-28 or 1-7* or decitabine IV on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  NOTE: Sonidegib PO QD is given on days 1-7 if in combination with azacitidine or on days 1-28 is given if in combination with decitabine.
  Interventions: Drug: Azacitidine; Drug: Decitabine; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Sonidegib

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Sonidegib — Given PO
  Other Names: ERISMODEGIB; LDE-225; LDE225; Odomzo; Smoothened Antagonist LDE225

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of azacitidine and sonidegib or decitabine and so see how well they work in treating patients with myeloid malignancies. The hedgehog (Hh) signaling pathway plays an important role in cellular growth, differentiation and repair. Inappropriate activation of Hh pathway signaling and uncontrolled cellular proliferation may be associated with mutations in the Hh-ligand cell surface receptor Smo. Sonidegib binds to the Hh cell surface receptor Smo, which may result in the suppression of the Hh signaling pathway and the inhibition of cancer cells. Azacitidine and decitabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving azacitidine together with sonidegib or decitabine may be a safe and successful treatment for patients with myeloid malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximally tolerated dose (MTD) of LDE225 (sonidegib) (days 1-28) in combination with azacitidine (overall); LDE225 (days 1-7) in combination with azacitidine (overall); and LDE225 (days 1-28) in combination with decitabine (overall). (Phase I) II. To estimate the efficacy of LDE225 (days 1-28) in combination with azacitidine in the following subgroups: untreated acute myeloid leukemia (AML)/chronic myelomonocytic leukemia (CMML)/myelodysplastic syndrome (MDS)/myeloproliferative neoplasm (MPN) overlap; relapsed/refractory AML/CMML/MDS/MPN overlap; and myelofibrosis (MF) only. (Phase Ib)

SECONDARY OBJECTIVES:

I. To estimate the duration of response, time to progression, overall survival, and time to AML or death (for MDS subjects) of LDE225 (days 1-28) in combination with azacitidine (overall and by cohort). (Phase I/1b)

TERTIARY OBJECTIVES:

I. To conduct correlative studies to measure HH pathway activation and inhibition and explore biomarkers of response.

II. To evaluate quality of life (QOL) and patient-reported symptoms using the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) and European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core (C)30 in subjects treated with LDE225 in combination with azacitidine or decitabine.

OUTLINE: This is a dose-escalation study of erismodegib.

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) on days 1-7, sonidegib orally (PO) once daily (QD) on days 1-28 or 1-7* or decitabine IV on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

*NOTE: Sonidegib PO QD is given on days 1-7 if in combination with azacitidine or on days 1-28 is given if in combination with decitabine.

After completion of study treatment, patients are followed up every 3 months until progressive disease and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of the following diagnoses:

  * Intermediate, high and very high risk (per International Prognostic Scoring System [IPSS]-revised [R]) untreated MDS or any MDS with >= 5% marrow blasts (by French American British [FAB] and World Health Organization [WHO] diagnostic criteria); NOTE: MDS/MPN overlap is allowed
  * CMML requiring treatment per doctor of medicine (MD) judgment
  * Low and very low risk MDS patients symptomatic and/or transfusion dependent, (>= 4 U red blood cells [RBC] over the preceding 12 week period) who have failed erythropoietin-stimulating agents (ESAs) or who have a low likelihood of responding to ESAs
  * MDS and CMML patients relapsed/refractory to hypomethylating agents as evidenced by one of the following:

    * Progressed at any time during treatment with hypomethylating agents
    * Failed to achieve a response after 6 cycles of 5-azacytidine or 4 cycles of decitabine
    * Progressed after treatment with hypomethylating agents had been discontinued

      * NOTE: MDS/MPN overlap is allowed
  * Relapsed or refractory AML exposed to =< 3 prior regimens (note, induction and consolidation including stem cell transplantation count as one regimen)
  * For exploratory phase I LDE225 days 1-7 with azacitidine or LDE225 days 1-28 with decitabine cohorts only: untreated AML/CMML/MDS/MPN overlap or relapsed/refractory AML/CMML/MDS/MPN overlap WITHOUT prior exposure to a hypomethylating agent (HMA)
  * Elderly (age >= 60) untreated AML and not a candidate for induction therapy
  * Untreated AML < 60 year of age who are not candidates to undergo standard induction chemotherapy
  * Primary myelofibrosis (PMF) and post essential thrombocytopenia (ET)/polycythemia vera (PV) MF with a Dynamic International Prognostic Scoring System (DIPSS)-plus score of intermediate or high, or a > 10% blasts in the marrow and who are in need of therapy and who have failed previous treatment with a janus kinase 2 (JAK2) inhibitor and, if appropriate, have failed Interferon based treatment
* Total bilirubin =< 1.5 mg/dL (except Gilbert's syndrome or known hemolysis or leukemic infiltration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x upper limit of normal (ULN) or < 5 x ULN if organ involvement
* Alkaline phosphatase < 5 x ULN
* Serum creatinine =< 1.5 x ULN or 24 hour creatinine (Cr) clearance > 50 ml/min
* Plasma creatine phosphokinase (CK) < 1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Ability to provide informed written consent and be able to adhere to the study visit schedule and other protocol requirements
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood and bone marrow aspirate samples for correlative research purposes
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Men must be willing to use appropriate contraception throughout study and for 6 months after; women must be willing to use appropriate contraception throughout study and for 20 months after
* Patients who have undergone stem cell transplantation (SCT), autologous or allogeneic, are eligible provided that they are > 84 days from stem cell infusion, have no active graft-versus-host disease (GVHD), are off immunosuppressive agents for > 14 days
* In the opinion of the investigator, patient must be able to receive at least 2 cycles of treatment

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection, known positive for active infectious hepatitis, type A, B or C; (past infection allowed), or psychiatric illness/social situations that would limit compliance with study requirements; Note: ongoing infection controlled on antibiotics/antifungal/antiviral medications are allowed unless listed as contraindicated
* Any of the following prior therapies:

  * Cytotoxic chemotherapy =< 14 days prior to registration
  * Immunotherapy =< 14 days prior to registration
  * Biologic therapy (i.e. antibody therapies) =< 14 days prior to registration
  * Radiation therapy =< 14 days prior to registration
  * Targeted therapies (i.e. kinase inhibitors, =< 7 days or 5 half-life's whichever is shorter)
  * Patients must be off other biologic therapies including hematopoietic growth factors >= 7 days prior to registration
  * For steroids or other non-cytotoxics given for blast count control, patient must be off for > 24 hours (hrs) before starting therapy; NOTE: hydroxyurea (HU) is allowed for blast count control throughout study
  * Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm =< 14 days prior to registration
* Active uncontrolled central nervous system (CNS) leukemia; NOTE: positive (cyto)pathology is allowed and patient can receive intrathecal chemotherapy
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Any previous treatment with LDE225 or allergic reactions to excipients of LDE225
* Acute promyelocytic leukemia (APL, M3) unless failed regimens that included tretinoin, arsenic trioxide, anthracyclines and cytarabine and currently NOT candidates for stem cell transplantation
* Major surgery =< 28 days prior to registration
* Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as 3-hydroxy-3-methylglutaryl-CoA (HMG CoA) inhibitors (statins), clofibrate and gemfibrozil, and that cannot be discontinued at least 5 half lives prior to starting LDE225 treatment; NOTE: if it is essential that the patient stays on a statin to control hyperlipidemia, only pravastatin may be used with extra caution
* Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment; NOTE: muscular activities, such as strenuous exercise, that can result in significant increases in plasma creatine kinase (CK) levels should be avoided whilst on LDE225 treatment
* Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)/cytochrome P450, family 3, subfamily A, polypeptide 5 (5) or drugs metabolized by cytochrome P450, family 2, subfamily B, polypeptide 6 (CYP2B6) or cytochrome P450, family 2, subfamily C, polypeptide 9 (CYP2C9) that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225; medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A4/5 inducers for at least 2 weeks prior to starting treatment with LDE225; NOTE: patients who are already on or require initiation of azoles other than fluconazole will be excluded from the phase I dose escalation portion of the study
* Impaired cardiac function or clinically significant heart disease, including any one of the following:

  * Angina pectoris within 3 months
  * Acute myocardial infarction within 3 months
  * Corrected Fridericia's QT (QTcF) > 450 msec for males and > 470 msec for females on the screening electrocardiogram (ECG)
  * A past medical history of clinically significant ECG abnormalities or a family history of prolonged QT-interval syndrome
  * New York Heart Association classification IV cardiovascular disease or symptomatic class III disease
  * Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception during the study and through 20 months after the final dose of study treatment if female, and for 6 months after final dose of study treatment if male
  * NOTE: adequate contraception is defined as either:

    * Total abstinence: when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Sterilization: patient has had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); (for female study patients, the vasectomized male partner should be the sole partner for that patient)
    * Use a combination of the following:

      * Placement of a non-hormonal intrauterine device (IUD) or non-hormonal intrauterine system (IUS)
      * Barrier method of contraception: condom or occlusive cap (diaphragm or cervical vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

        * Note: hormonal contraception methods (e.g. oral, injected, implanted) are not allowed as it cannot be ruled out that the study drug decreases the effectiveness of hormonal contraception
        * Note: women are considered post-menopausal and not child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
        * Note: male patient must use highly effective (double barrier) methods of contraception (e.g., spermicidal gel plus condom) for the entire duration of the study, and continuing using contraception and refrain from fathering a child for 6 months following the study drug; a condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the study treatment via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Best overall response (complete response [CR] or complete response with incomplete recovery [CRi]) in untreated AML, CMML, MDS, or MDS/MPN Overlap patients (Phase IB [Dose Expansion]) | Up to 30 days post-treatment
  The proportion of CR/CRi responses will be estimated (by cohort) by the number of CR/CRi responses divided by the total number of evaluable patients. 95% exact binomial confidence intervals will be computed. The frequency and relative frequency of individual response categories will also be computed. Best overall response over all cycles of study treatment will also be described using frequency and relative frequency of individual response categories.
Best overall response (CR or CRi) in myelofibrosis patients (Phase IB [Dose Expansion]) | Up to 30 days post-treatment
  The proportion of CR/CRi responses will be estimated (by cohort) by the number of CR/CRi responses divided by the total number of evaluable patients. 95% exact binomial confidence intervals will be computed. The frequency and relative frequency of individual response categories will also be computed. Best overall response over all cycles of study treatment will also be described using frequency and relative frequency of individual response categories.
Best overall response (CR or CRi) in relapsed/refractory AML, CMML, MDS, or MDS/MPN Overlap patients (Phase IB [Dose Expansion]) | Up to 30 days post-treatment
  The proportion of CR/CRi responses will be estimated (by cohort) by the number of CR/CRi responses divided by the total number of evaluable patients. 95% exact binomial confidence intervals will be computed. The frequency and relative frequency of individual response categories will also be computed. Best overall response over all cycles of study treatment will also be described using frequency and relative frequency of individual response categories.
MTD defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) (Phase I) | 42 days
  Graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.

SECONDARY OUTCOMES:
Duration of response | Date at which the patient's earliest best objective status is first noted to be a CR/CRi response to the earliest date progression is documented, assessed up to 30 days post-treatment
  The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Incidence of adverse events graded using the NCI CTCAE version 4.0 (Phase IB [dose expansion]) | Up to 30 days post-treatment
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns (by cohort and overall). Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. The rate of grade 3 or higher non-hematologic adverse events, and the rate of grade 4 or higher adverse event (hematologic and non-hematologic) will be computed each with a 95% exact binomial confidence interval.
Overall survival | Time from registration to death due to any cause, assessed up to 30 days post-treatment
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to AML | Time from registration to leukemic transformation due to any cause, assessed up to 30 days post-treatment
  The distribution of time to AML will be estimated using the method of Kaplan-Meier.
Time to death | Time from registration to death due to any cause, assessed up to 30 days post-treatment
  The distribution of time to death will be estimated using the method of Kaplan-Meier.
Time to progression | Time from registration to the earliest date of documentation of disease progression, assessed up to 30 days post-treatment
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.

OTHER OUTCOMES:
Biomarker levels | Up to 30 days post-treatment
  Statistical analysis of each biomarker will be primarily descriptive. Continuous biomarker levels will be explored in a graphical manner including mean plots and plots of change and percent change from baseline and other summary measures. Any potential relationships between the baseline level or change in the level of each biomarker and clinical outcome such as overall response, 6-month progression and survival, and adverse event incidence will be further analyzed using Wilcoxon rank sum tests or logistic regression methods, as appropriate.
Patient-reported outcomes (quality of life and symptoms) as assessed by the EORTC QLQ-C30 and MPN-SAF Total Symptom Score (TSS) | Up to 30 days post-treatment
  Scale score trajectories over time will be examined using stream plots and mean plots with standard deviation error bars overall. Changes from baseline at each cycle will be statistically tested using paired t-tests, and standardized response means (mean of the change from baseline scores at a given cycle, divided by the standard deviation of the change scores) will be interpreted (after applying Middel's adjustment) using Cohen's cut-offs.

CONTACTS AND LOCATIONS:
Overall Officials: Aref Al-Kali, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials